CLINICAL TRIAL: NCT06832644
Title: Novel Risk Prediction Approaches for the Primary Prevention of Cardiovascular Diseases in Italy: the CVRISK-IT Trial
Brief Title: Novel Risk Prediction Approaches for the Primary Prevention of Cardiovascular Diseases in Italy: the CVRISK-IT Trial (CVRISK-IT)
Acronym: CVRISK-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Centro Cardiologico Monzino (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Istituti Clinici Scientifici Maugeri SpA (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); IRCCS Multimedica (Other); Istituto Neurologico Mediterraneo Neuromed S. R. L (Other); IRCCS San Raffaele (Other); IRCCS San Raffaele Roma (Other); IRCCS SYNLAB SDN (Other); Istituto Clinico Humanitas (Other); Istituto Nazionale di Ricovero e Cura per Anziani (Other); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Ospedale Policlinico San Martino (Other); Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Lorenzo Menicanti, MD, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CVRISK-IT
Record Dates: First submitted 2025-02-04; First posted 2025-02-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Risk; Genetic Cardiovascular Risk
Keywords: Primary Prevention; Cardiovascular Risk; SCORE2/2-OP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No additional cardiovascular risk information/recommendation is provided to the subject other than SCORE2/SCORE2-OP results of phase I. Thereby, the control group does not undergo neither imaging nor genetic analysis.
- Imaging (Experimental): Subjects randomized in the imaging arm receive personalized recommendations on lifestyle and, if necessary, therapeutic intervention based on imaging data analysis (i.e., carotid ultrasound or calcium score)
  Interventions: Behavioral: Lifestyle Management
- Polygenic Risk Score (PRS) (Experimental): Subjects randomized in this arm receive personalized recommendations on lifestyle and, if necessary, therapeutic intervention based on polygenic risk score (PRS) analysis obtained from blood samples collected at the baseline visit
  Interventions: Behavioral: Lifestyle Management
- Imaging and Polygenic Risk Score (PRS) (Experimental): Subjects randomized in this arm receive personalized recommendations on lifestyle and, if necessary, therapeutic intervention based on both imaging data (e.g., carotid ultrasound and/or calcium score) and genetic analysis (e.g., PRS).
  Interventions: Behavioral: Lifestyle Management

INTERVENTIONS:
Behavioral: Lifestyle Management — All individuals will receive tailored lifestyle advice along with medical treatment based on their newly estimated CVD risk. The control group will also receive lifestyle advice along with medical treatment based only on their CVD risk provided at the baseline visit during phase I.
  Arms: Imaging; Imaging and Polygenic Risk Score (PRS); Polygenic Risk Score (PRS)

SUMMARY:
The CVRISK-IT study aims to evaluate the health benefit of measuring genetic and imaging risk information in men and women considered at 'low-to-moderate' or 'high' risk of developing cardiovascular diseases (CVD) in a randomized controlled trial in Italian primary care settings. Our primary objective is to answer a fundamental question in the prevention and prediction of CVD in Italy and globally: is there any benefit in including additional information (such as genetic and/or imaging data) in estimating risk, in conjunction with lifestyle advice and medical treatment for primary prevention of CVD?

As a key secondary objective of the CVRISK-IT study, the goal is to build a large bioresource with clinical information and biological samples to facilitate a new generation of discovery and translational research that will advance understanding of the genetic, molecular and behavioural determinants as well as mechanisms of multiple chronic diseases in the Italian population. By contributing to the Rete Cardiologica database and the BBDCARDIO biobank, the CVRISK-IT study will also serve as a cornerstone for future investigations into the development and testing of early diagnostic technologies and preventive (or 'personalised precision health') interventions for chronic diseases.

DETAILED DESCRIPTION:
This multicenter, open randomized trial will investigate the effects of providing additional CVD risk information alongside personalised lifestyle advice and medical treatment in a primary prevention context across Italy. Healthy individuals aged 40 to 80 years, with no prior history of CVD or diabetes, will be recruited in two phases from the cohort of 17 participating IRCCS across Italy and affiliated enrolling centers. The population enrolled in this study consists of subjects who have never participated in other cardiovascular prevention studies of the Rete Cardiologica.

Phase 1 - Identification of the study population and development of the bioresource: various recruitment sources will be used, including institutions, primary care centres/services, government agencies, occupational health services, and volunteer organizations (e.g., blood donors). Participants will provide informed consent, a blood sample, and complete an electronic questionnaire. Approximately 30,000 individuals will be recruited and assessed using SCORE2/SCORE2-OP risk prediction models. Those identified as 'very high' risk will receive immediate medical treatment and will not proceed to phase 2.

Phase 2 - Randomization and novel risk prediction interventions: Participants identified as 'low-to-moderate' or 'high' CVD risk during phase 1 will be randomized, following a 2x2 factorial design into four groups within 1 week upon enrolment: a control group (no additional risk information), and three intervention groups (genetic, imaging-based and genetic + imaging-based risk information). The goal is to randomize around 12,000 participants in phase 2 (~3,000 per trial arm). All individuals will receive tailored lifestyle advice along with medical treatment based on their newly estimated CVD risk. The remaining 18,000 participants who won't proceed to phase 2 will still be involved in the study and contacted through a phone call follow-up with specialist at the 5◦ and 10◦ year.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-80 years
* Apparently healthy individuals without previous medical history of CVD or diabetes (based on medical diagnosis)
* Participant recruitment arranged only at selected IRCCS (and associated Spokes) as part of the 'Rete Cardiologica'
* Participants must have signed the Informed Consent and Data Privacy Treatment forms
* Participants must have a personal e-mail address and internet connection

Exclusion Criteria:

* Age ≤40 or ≥80 years
* Individuals have previous medical history related to CVD (e.g., heart failure, congenital heart disorder, coronary heart disease) based on medical diagnosis
* Candidates have previously participated in clinical studies of 'Rete Cardiologica' (e.g., PREVITAL)
* Medical diagnosis of mental disorders
* Pregnancy based on self-reported information
* Previous history of type 1 or type 2 diabetes (based on medical diagnosis)
* Oncology patients (based on physician indication)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30000 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in CVD risk using SCORE2/SCORE2-OP | 12 months
  The primary short-term outcome (i.e., 12 months after communication of the newly estimated CVD risk, following the randomisation step) is the change in CVD risk measured using SCORE2/SCORE2-OP risk prediction models. The CVD risk categories used to classify healthy people according to these scores are: 1) Low-to-moderate CVD risk: <50 years = <2.5 %; 50-69 years = <5%; ≥ 70 years = <7.5%. High CVD risk: <50 years = 2.5 to <7.5%; 50-69 years = 5 to <10%; ≥ 70 years 7.5 to <15%; Very high CVD risk: <50 years = ≥7.5%; 50-69 years = ≥10%; ≥ 70 years = ≥ 15%.

SECONDARY OUTCOMES:
Change in cardiovascular modifiable risk factors | 12 months
  Secondary short-term outcomes will include changes in objectively measured risk factors, such as cholesterol levels (i.e., total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides) (mg/dl)
Change in cardiovascular modifiable risk factors | 12 months
  Secondary short-term outcomes will include changes in objectively measured risk factors, such as blood pressure which will be measured 3 times in a row, and its average calculated (mmHg)
Change in cardiovascular modifiable risk factors | 12 months
  Secondary short-term outcomes will include changes in objectively measured risk factors, such as smoking habits (e.g., switch from "usual smoker" to "not smoking anymore" categories)
Change in CVD prevention-drugs prescription | 12 months
  Secondary short-term outcomes will include changes in CVD prevention-drugs prescription with respect to the baseline visit
Evaluation of participant's adherence to ESC recommendations | 12 months
  By means of validated questionnaires, the assessment of participants' adherence to the lifestyle and dietary guidelines of the European Society of Cardiology (ESC) will be performed. If and where applicable, drugs prescription adherence will be evaluated as well as psychological outcomes

OTHER OUTCOMES:
CVD events recording in long-term period | 5-10 years
  The long-term outcomes will include the registration of CVD events in all enrolled participants in the long-term period (e.g., non-fatal myocardial infarction, acute coronary syndrome, percutaneous transluminal coronary angioplasty (PTCA), Coronary artery bypass grafting (CABG), non-fatal stroke), CVD mortality, and total mortality

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (17):
  - IRCCS Cardiologico Monzino, Milan, Milan
  - Irccs Inrca, Ancona
  - IRCCS San Martino, Genova
  - IRCCS Auxologico Italiano, Milan
  - IRCCS Fondazione Cà Granda- Policlinico Milano, Milan
  - IRCCS Istituto Clinico Humanitas, Milan
  - IRCCS Mario Negri, Milan
  - IRCCS Multimedica, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Irccs Synlab Sdn, Naples
  - Irccs Ismett, Palermo
  - IRCCS Fondazione Policlinico San Matteo, Pavia
  - IRCCS Istituti Clinici Scientifici Maugeri, Pavia
  - IRCCS Neuromed, Pozzilli
  - IRCCS Fondazione Policlinico Gemelli, Rome
  - IRCCS San Raffaele Roma, Rome
  - IRCCS Policlinico San Donato, San Donato Milanese

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Timmis A, Vardas P, Townsend N, Torbica A, Katus H, De Smedt D, Gale CP, Maggioni AP, Petersen SE, Huculeci R, Kazakiewicz D, de Benito Rubio V, Ignatiuk B, Raisi-Estabragh Z, Pawlak A, Karagiannidis E, Treskes R, Gaita D, Beltrame JF, McConnachie A, Bardinet I, Graham I, Flather M, Elliott P, Mossialos EA, Weidinger F, Achenbach S; Atlas Writing Group, European Society of Cardiology. European Society of Cardiology: cardiovascular disease statistics 2021. Eur Heart J. 2022 Feb 22;43(8):716-799. doi: 10.1093/eurheartj/ehab892. PMID 35016208